CLINICAL TRIAL: NCT00960557
Title: A Multicenter, Open-label Phase 1b/2 Study to Assess the Safety and Clinical Activity of Intravenous Combretastatin A1 Diphosphate (OXi4503) as Monotherapy in Subjects With Primary or Secondary Hepatic Tumor Burden
Brief Title: Safety Study of Increasing Doses of Combretasatin A1 Diphosphate (OXi4503) as Monotherapy in Subjects With Hepatic Tumor Burden
Acronym: OXi4503
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mateon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OXC101-100
Record Dates: First submitted 2009-08-14; First posted 2009-08-18 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Neoplasm Metastasis
Keywords: hepatic tumor burden; liver cancer; liver carcinoma; carcinoma; hepatic cancer; hepatic carcinoma; VDA; Vascular Disrupting Agent
MeSH Terms: conditions — Neoplasm Metastasis; Liver Neoplasms; Carcinoma, Hepatocellular; Carcinoma | interventions — Oxi 4503

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combretastatin A1 Diphosphate (Experimental)
  Interventions: Drug: Combretastatin A1 Diphosphate (OXi4503)

INTERVENTIONS:
Drug: Combretastatin A1 Diphosphate (OXi4503) — OXi4503 administered IV on Days 1, 8, and 15 of each 28-day cycle.

SUMMARY:
The purpose of this study is to determine the safety and tolerability of OXi4503 in subjects with relapsed or refractory carcinomas with hepatic tumor burden.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed carcinoma. Tumor must be relapsed or refractory to standard therapies, or have no acceptable standard therapy.
2. Measurable disease by RECIST criteria.
3. Subjects must be at least 28 days from other investigational therapy and at least 2 weeks after chemotherapy or radiation therapy.
4. Age 18 years or older.
5. Eastern Cooperative Oncology Group (ECOG) Performance Score of less than 1.
6. Life expectancy of greater than 12 weeks.
7. Hemoglobin greater than 10 g/dL.
8. Adequate hepatic function.
9. Adequate renal function.
10. Adequate bone marrow reserve.
11. Able to maintain potassium, calcium and magnesium levels within normal ranges.
12. Must be able to provide written informed consent.
13. All women of childbearing potential (WOCBP) must have a negative serum pregnancy test.
14. WOCBP and fertile men and their partners must agree to use an effective form of contraception during the study and for 90 days after the last dose of study medication.

Exclusion Criteria:

1. Uncontrolled CNS metastases.
2. No other active malignancies.
3. Poorly controlled hypertension.
4. Recent history of serious cardiovascular conditions.
5. Recent history of CVA, TIA, or intermittent claudication.
6. Current anticoagulation therapy.
7. History of cardiac arrhythmias.
8. Abnormal ECG findings.
9. Subjects who require concomitant medications which cause QTc prolongation.
10. Major surgery within 30 days of treatment, or minor surgery within 7 days of treatment.
11. Uncontrolled, clinically significant active infection.
12. Subjects who are pregnant or lactating.
13. Subjects with any other intercurrent medical condition.
14. Subjects with a history of solid organ transplant or bone marrow transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of OXi4503 in subjects with relapsed or refractory carcinomas with hepatic tumor burden. | 6 Months

SECONDARY OUTCOMES:
To determine progression-free survival (PFS). | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Brown, MD, Principal Investigator — Royal Adelaide Hospital; Jason Lickliter, MD, Principal Investigator — Monash Medical Centre; Paul Mainwaring, MD, Principal Investigator — Mater Adult Hospital; Michael Millward, MD, Principal Investigator — Sir Charles Gairdner Hospital
Locations (4):
- Australia (4):
  - OXiGENE Investigational Site, Westmead, New South Wales
  - OXiGENE Investigational Site, South Brisbane, Queensland
  - OXiGENE Investigational Site, Adelaide, South Australia
  - OXiGENE Investigational Site, Bentleigh, Victoria

REFERENCES:
- [Derived] Giri P, Batra PJ, Kumari A, Hura N, Adhikary R, Acharya A, Guchhait SK, Panda D. Development of QTMP: A promising anticancer agent through NP-Privileged Motif-Driven structural modulation. Bioorg Med Chem. 2023 Nov 15;95:117489. doi: 10.1016/j.bmc.2023.117489. Epub 2023 Oct 5. PMID 37816266